CLINICAL TRIAL: NCT03128398
Title: Use of Domperidone for Treatment of Upper Gastrointestinal Disorders
Acronym: Domperidone
Status: No longer available | Type: Expanded Access
Sponsor: Palo Alto Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PACR-14-04-311
Record Dates: First submitted 2017-04-06; First posted 2017-04-25 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Gastroparesis
Keywords: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Domperidone

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Domperidone — Availability of Domperidone to patients with serious gastrointestinal diseases or conditions when there is no comparable or satisfactory alternative therapy to diagnose, monitor, or treat the patient's disease or condition.

SUMMARY:
This is an Expanded Access to Investigational Drug program available through the FDA. Some specific conditions to qualify for this program includes gastroesophageal reflux disease with upper GI symptoms, gastroparesis, and chronic constipation. Patients failing standard therapies for these conditions may be eligible to receive domperidone. This program facilitates availability of investigational drugs, (such as domperidone) to patients with serious diseases or conditions when there is no comparable or satisfactory alternative therapy to diagnose, monitor or treat the patients's disease or condition. Authorization must be obtained from FDA prior to the importation, interstate shipment and administration of domperidone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 18 and older
3. Symptoms or manifestations secondary to motility disorders of the upper GI tract. These include gastroparesis, functional dyspepsia, gastroesophageal reflux disease that are refractory to standard therapy.
4. Patients must have a comprehensive evaluation to eliminate other causes of their symptoms. This includes a history and physical examination. A recent (within 3 years) evaluation of the upper GI tract with either upper endoscopy or upper GI radiographic series. Baseline blood tests suggested are electrolytes, magnesium, and prolactin level.
5. Patient has signed informed consent for the administration of domperidone that informs the patient of potential adverse events including:

   * Increased prolactin levels
   * Breast changes
   * Extrapyramidal side effects
   * Cardiac arrhythmias including QT prolongation (increased risk with the drugs listed in the appendix)

Exclusion Criteria:

History of, or current, arrhythmias including ventricular tachycardia, ventricular fibrillation and Torsade des Pointes. Patients with minor forms of ectopy (PACs) are not necessarily excluded.

2. Clinically significant bradycardia, sinus node dysfunction, or heart block. Prolonged QTc (QTc > 450 milliseconds for males, QTc > 470 milliseconds for females).

3. Clinically significant electrolyte disorders. These include significant hypokalemia, hyperkalemia, hypomagnesemia, and hypermagnesemia that cannot be corrected with treatment of these electrolyte abnormalities.

4. Gastrointestinal hemorrhage or obstruction. 5. Presence of a prolactinoma (prolactin-releasing pituitary tumor). 6. Pregnant or breast feedings female. 7. Known allergy to domperidone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Shetler, MD, Principal Investigator — Palo Alto Medical Foundation